CLINICAL TRIAL: NCT02276183
Title: Effects of a Test Formula Milk Powder Combined With a Physical Activity Program on Mobility in Healthy Aging Subjects With Joint Discomfort
Brief Title: Move Study in Healthy Aging People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13.25 NRC
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm1, Nutrition intervention, test formula and activity (Experimental)
  Interventions: Dietary Supplement: Nutrition intervention, test formula; Behavioral: progressive physical activity

INTERVENTIONS:
Dietary Supplement: Nutrition intervention, test formula
Behavioral: progressive physical activity — Tai Chi; dynamic strength training (knee extension, knee flexion, hip extension, side leg raise, plantar flexion); flexibility warm up and cool down (shoulder and upper arm stretch, hamstrings stretch, calf stretch, ankle stretch); aerobic fitness training(walking on even flat ground); balance training(standing on one foot; heel-to-toe walk; toe stand)

SUMMARY:
Bone and muscle losses occur during ageing leading to increased risk of osteoporosis (there are more than 200 million people affected by osteoporosis worldwide), sarcopenia, loss of functionality and mobility. From around 45-50 years onwards, there is a progressive loss of muscle mass and strength (sarcopenia). This is partially due to an impairment of muscle protein synthesis in response to dietary proteins. Insufficient dietary protein may contribute to age-related loss of lean body mass (LBM) and strength which ultimately affects body movement.

Key ingredients in selected investigational product are:Milk proteins, Calcium, Vitamin D, Vitamin C, Glucosamine Sulfate, Zinc. They have effects to improve physical mobility and functionality. The investigators expect improved effects of a nutritional intervention combined with a physical activity program on mobility in healthy aging subjects with joint discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Target 45-65 y old
* Suffering from (knee) pain. VAS on pain assessment <= 4 on a range 0 to 10
* 20<BMI<28
* Time since menopause above 2y
* iPAQ (International Physical Activity Questionnaire) score <600

Exclusion Criteria:

* OA diagnosed
* Medicine treatment
* Chronic pain killers treatment for more than 7 consecutive days with a washout period of 2 weeks between 2 periods of treatment
* Under corticoid, hormone (adrenal, thyroid) treatment
* Traditional herbal medicine: in particular with claims on strengthening tendons and bones. This point will be included in FFQ (see annex) and evaluate.

Subjects with chronic tablets supplementation ( calcium or drinking milk over 5 day wk-1 will be excluded, vitamin D, GS, or any with effect on bone and joints ) (set up a FFQ to specially investigate intakes of calcium tablets, milk and animal foods)

* Pregnancy
* Subject with knee/joint surgery/replacement and CLA (Cross Ligament) injury
* History of relevant digestive disease, organic disease of heart, liver or kidney, severe function disorder of liver or kidney, metabolic/endocrine , neurological disease (e.g., Parkinson disease, stroke) with residual impairment, vertigo
* Anaemia
* Unable to carry out functional tests and questionnaires correctly (KOOS, physical activity)
* Lower or upper extremity surgery or fracture in the last 3 months
* Currently participating or having participated in another clinical trial in the three previous months

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in muscle extension isokinetic strength and 4 min speed step | Baseline and visit 7
  Change from baseline and muscle(quadriceps)extension isokinetic strength (peak torque) and 4 min speed step will be measured as the change of musculoskeletal functionality and mobitliy.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China